CLINICAL TRIAL: NCT04615962
Title: A Phase I, Multicenter, Double-Blind, Randomized Study to Evaluate the Safety and Tolerability Profile of Topical Cream SNG100 for 14 Days of Treatment in Moderate Atopic Dermatitis Subjects.
Brief Title: Topical Cream SNG100 for Treatment in Moderate Atopic Dermatitis Subjects.
Acronym: SNG100
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seanergy Dermatology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CSP-001-SNG1
Record Dates: First submitted 2020-10-25; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — hydrocortisone acetate; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SNG100 (Experimental): Combination of low potency steroid with hydrating and moisturizing agents
  Interventions: Drug: SNG100
- Hydrocortisone (Active Comparator): This medication is used to treat a variety of skin conditions (e.g., eczema, dermatitis, allergies, rash).
  Interventions: Drug: Hydrocortisone Acetate 1% Cream
- Mometasone furoate (Active Comparator): This medication is used to treat skin conditions such as eczema, psoriasis, allergies, and rash.
  Interventions: Drug: Mometasone Furoate

INTERVENTIONS:
Drug: Hydrocortisone Acetate 1% Cream — Hydrocortisone Acetate is the synthetic acetate ester form of hydrocortisone, a corticosteroid with anti-inflammatory and immunosuppressive properties.
  Arms: Hydrocortisone
Drug: Mometasone Furoate — Mometasone is a medium-strength corticosteroid.
  Arms: Mometasone furoate
Drug: SNG100 — A combination of low potency steroid and skin barrier repair agent
  Arms: SNG100

SUMMARY:
The investigators aimed to understand better the efficacy in a randomized, double-blind, intraindividual design trial in 66 participants with AD treated with SNG100, and 2 different strengths of topical steroids hydrocortisone and the medium potent mometasone furoate cream.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 6 years old or older with a diagnosis of moderate atopic dermatitis confirmed by a dermatologist
2. Any child age 6 to 18 with a diagnosis of moderate atopic dermatitis confirmed by a dermatologist, together with the child's parent/guardian. Written informed consent must be given by parent/guardian.
3. Capable of complying with study requirements and study procedure.
4. Investigator Global Assessment (IGA) of 3.
5. The severity of atopic dermatitis will be defined as moderate by SCORAD range of 26-50 and EASI range of 7.1-21 points.
6. Child-bearing potential women must use a proper contraception method.

Exclusion Criteria:

1. As determined by the study doctor, a medical history that may interfere with study objectives.
2. Atopic dermatitis lesions that occur only on the face and scalp.
3. Presence of a secondary infection with bacteria, fungi, or virus.
4. Recent or current participation in another research study.
5. Females who are breastfeeding, pregnant, or with plans to get pregnant during the participation in the study.
6. Prior wound, tattoo, pigmentation or infection in the treated area.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Side Effects AE's and SAE's | 4 weeks
  Evaluate safety and tolerability as measured by completion of a full prescribed treatment course, treatment interruptions, SAE's and AE's

SECONDARY OUTCOMES:
Usability | 4 weeks
  Within subject difference in response to topical product usability questionnaire items between trial treatments

OTHER OUTCOMES:
Change from baseline in the SCORAD index | 4 weeks
  SCORAD: SCOring of Atopic Dermatitis
  Subscales:
  Eczema Spread (A): 0 - 20 Eczema Intensity (B): 0 - 63 Subjective Symptoms (C): 0 - 20 Total = (A/5) + (Bx7/2) + C Total: 0 - 103 (Higher values represent a worse outcome)
Eczema Area and Severity Index (EASI) Score | 4 weeks
  The surface and severity of eczema is measured using the Eczema Area and Severity Index (EASI). A regional body surface area tabulation based on severity ranging from 0 (none) to 3 (severe), and severity of signs of disease, then multiplied by body area with final possible calculation ranging from 0 (none) - 72 (severe).
NRS score | 4 weeks
  Itch Numeric Rating Scale. 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity.
Investigator's Global Assessment (IGA) Score | 4 weeks
  The IGA measures the investigator's global assessment of the participants overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Ramot, Prof., Study Director — Seanergy Ltd.

IPD SHARING:
Plan to Share IPD: No